CLINICAL TRIAL: NCT01018862
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-36 (0.15% Solution) and MP03-33 (0.10% Solution) in Children Ages >6 to <12 With Perennial Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Efficacy of a Nasal Spray to Treat Children With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP441
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-05

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MP03-36 (0.15% solution) (Active Comparator): 822 mcg, Topical/intranasal spray, 1 spray per nostril twice daily/ 4 weeks
  Interventions: Drug: Azelastine hydrochloride nasal spray 0.15%
- MP03-33 (0.10% solution) (Active Comparator): 548 mcg, Topical/intranasal spray, 1 spray per nostril twice daily/ 4 weeks
  Interventions: Drug: Azelastine hydrochloride nasal spray 0.10%
- Placebo (Placebo Comparator): 0 mcg, Topical/intranasal spray, 1 spray per nostril twice daily/ 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azelastine hydrochloride nasal spray 0.15% — 822 mcg, Topical/intranasal spray, 1 spray per nostril twice daily/ 4 weeks
  Other Names: Astepro 0.15%
  Arms: MP03-36 (0.15% solution)
Drug: Azelastine hydrochloride nasal spray 0.10% — 548 mcg, Topical/intranasal spray, 1 spray per nostril twice daily/ 4 weeks
  Other Names: Astepro 0.10%
  Arms: MP03-33 (0.10% solution)
Drug: Placebo — 0 mcg, Topical/intranasal spray, 1 spray per nostril twice daily/ 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness of an Investigational use of an allergy medication (MP03-33) used to treat perennial allergic rhinitis (PAR) to placebo (a nasal spray that contains no medicine). In addition, the study will also compare the safety and effectiveness of an investigational use of another allergy medication (MP03-36) used to treat perennial allergic rhinitis to placebo.

DETAILED DESCRIPTION:
in Children Ages >6 to <12 with Perennial Allergic Rhinitis (PAR)

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects >6-<12, inclusive at the screening visit
* At least a 1-year history of PAR
* The parent must provide written informed consent and the child must provide written assent.
* Willing and able to comply with the study requirements
* The presence of immunoglobulin E (IgE)-mediated hypersensitivity to dust mite, cockroach, mold, cat or dog dander, confirmed by a positive response to skin prick testing at the Visit 1. A positive response is defined as a wheal diameter of ≥5 mm larger than the negative control for the skin prick test. Histamine control must also be positive with a wheal diameter >5 mm larger than the control. If there are prevailing seasonal allergies, the subject must have a negative skin test to the specific allergen.
* Screening Visit: Have a 12-hour reflective TNSS of at least 6 out of a possible 12 and a congestion score of ≥2 or a rhinorrhea score of ≥2 on Visit 1
* Randomization Visit: to be eligible for entry into the double-blind treatment period, subjects/caregivers must record:

  1. at least 3 symptom assessments (either AM or PM score) during the past 3 days of the Lead-In Period or the Day of Randomization:

     1. a 12-hour reflective TNSS ≥ 6
     2. a 12-hour reflective congestion score of ≥2 or a rhinorrhea score of ≥2
  2. the total of the seven Lead-In symptom assessments during the past 3 days of the Lead-In Period including the Day of Randomization (Visit 2/Day 1):

     1. a 12-hour reflective TNSS ≥ 42
     2. a 12-hour reflective congestion score of ≥14 or a rhinorrhea score of ≥14
* Must have taken at least 10 doses of study medication during the placebo Lead-In Period
* General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
* Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections do not preclude participation). Subjects receiving sublingual immunotherapy are excluded. A 6 month washout period is required following the last dose of sublingual immunotherapy.

Exclusion Criteria:

* On nasal examination, subjects with superficial nasal mucosal erosion, moderate nasal mucosal erosion, nasal mucosal ulceration, nasal septum perforation (Grade 1B - 4) (see section 8.1.4).
* Other nasal disease(s) likely to affect deposition of intranasal medication, such as acute sinusitis, rhinitis medicamentosa or clinically significant polyposis or nasal structural abnormalities.
* Nasal surgery or sinus surgery within the previous year.
* Chronic sinusitis
* The use of any investigational drug within 30 days prior to Visit 1. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
* Females who are pregnant or nursing
* Females of childbearing potential who are not abstinent and not practicing a medically acceptable method of contraception
* Respiratory tract infections within two weeks prior to Visit 1
* Subjects with significant pulmonary disease including asthma. Subjects with intermittent asthma who only require short-acting inhaled bronchodilators are eligible for enrollment.
* Chronic obstructive sleep apnea syndrome (clinical diagnosis)
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug or that might significantly affect the subject's ability to complete this trial.
* Clinically relevant abnormal physical findings within 1 week of randomization which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures
* Overnight absences from home for more than 3 nights
* Family members of research center or private practice personnel who are directly involved in this study are excluded
* Members of the same family cannot enroll in the study at the same time
* Subjects who have used the medications or therapies that could interfere with symptom evaluation within the time period specified (see Section 4.0).
* Any behavioral condition which could affect subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 489 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ginsberg, DO, Study Director — Meda Phamaceuticals, Sr.Dir Medical and Scientific Affairs
Locations (39):
- United States (39):
  - West Coast Clinical Trials, Costa Mesa, California
  - Allergy, Asthma and Respiratory Care Center, Long Beach, California
  - Southern California Research, Mission Viejo, California
  - Joann Blessing-Moore,MD, Palo Alto, California
  - Capital Allergy and Respiratory Disease Center, Sacramento, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Cntr, San Jose, California
  - Bensch Research Associates, Stockton, California
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Center for Allergy, Asthma and Immunology, Waterbury, Connecticut
  - Clinical Research Atlanta, Atlanta, Georgia
  - Idaho Allergy, Eagle, Idaho
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Clinical Research Institute of Indiana, Indianapolis, Indiana
  - Chesapeake Clinical Research, Inc, Baltimore, Maryland
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - Clinical Research Institute, Plymouth, Minnesota
  - Asthma and Allergy Center, PC, Papillion, Nebraska
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Asthma, Sinus & Allergy Centers, LLC, Warren Township, New Jersey
  - Island Medical Research, Rockville Centre, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy and Asthma, Oklahoma City, Oklahoma
  - Baker Asthma, Allergy and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Allergy Associated Research Center, Portland, Oregon
  - Allergy and Asthma Consultants of NJ-PA, P.C, Collegeville, Pennsylvania
  - Allergy and Asthma Consultants, LLP, Charleston, South Carolina
  - Isis Clinical Research, LLC, Ausitn, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Sirius Clinical Research, Austin, Texas
  - Pharmaceutical Research & Consulting Inc, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Marycliff Allergy Specialists, Spokane, Washington
  - Gary Steven, MD, Greenfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo
Started | 161 | 166 | 162
Completed | 148 | 156 | 146
Not Completed | 13 | 10 | 16
Not completed — Adverse Event | 2 | 0 | 6
Not completed — Lack of Efficacy | 1 | 0 | 2
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Protocol Violation | 1 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — administrative problems | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo | Total
Number analyzed (Participants) | 161 | 166 | 162 | 489
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 161 | 166 | 162 | 489
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.8 (2.6) | 8.8 (2.7) | 8.7 (2.8) | 8.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 65 | 69 | 208
  Male | 87 | 101 | 93 | 281
Region of Enrollment [Number; unit: participants]
  United States | 161 | 166 | 162 | 489

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score (TNSS) for the Entire 28-day Study Period Compared to Placebo
Description: Change from baseline in 12-hour reflective total nasal symptom score (TNSS) for the entire 28-day study period compared to placebo,scored on a 0 to 24 scale with 0 being no symptoms and 24 being severe symptoms.
Time Frame: baseline to 28 Days
Population: participant must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo
Number analyzed (Participants) | 159 | 166 | 161
units on a scale | -3.45 (4.03) | -3.37 (4.37) | -2.48 (3.93)

2. Secondary Outcome: Change From Baseline in the Instantaneous Total Nasal Symptoms Score (TNSS) for the Entire 28-day Study Period Compared to Placebo
Description: change from baseline in 12-hour instantaneous total nasal symptom score (TNSS) for the entire 28-day study period compared to placebo,scored on a 0 to 24 scale with 0 being no symptoms and 24 being severe symptoms.
Time Frame: baseline to 28 days
Population: participant must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo
Number analyzed (Participants) | 159 | 165 | 161
units on a scale | -2.70 (3.91) | -3.00 (4.42) | -2.38 (3.95)

3. Secondary Outcome: Change From Baseline in 12-hour Reflective Total Ocular Symptoms Score (TOSS) and Instantaneous Total Ocular Symptoms Score (TOSS) for the Entire 28-day Study Period Compared to Placebo
Description: change from baseline in 12-hour instantaneous total ocular symptom score (TOSS) for the entire 28-day study period compared to placebo,scored on a 0 to 18 scale with 0 being no symptoms and 18 being severe symptoms.
Time Frame: baseline to 28 days
Population: participant must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo
Number analyzed (Participants) | 157 | 164 | 160
units on a scale | -1.46 (2.72) | -1.51 (3.12) | -1.28 (3.01)

4. Secondary Outcome: Change From Baseline to Visit 4 in the Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Compared to Placebo
Description: change from baseline in the Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) compared to placebo for the entire 28-day study period compared to placebo,scored on a 0 to 42 scale with 0 being not troubled at all and 42 being extremely troublesome.
Time Frame: baseline to 28 Days
Population: participant must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo
Number analyzed (Participants) | 158 | 164 | 160
units on a scale | -0.30 (0.95) | -0.38 (0.87) | -0.38 (0.83)

ADVERSE EVENTS:
Arm/Group | MP03-36 (0.15% Solution) | MP03-33 (0.10% Solution) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/166 | 0/162
Other Adverse Events (participants affected / at risk) | 39/161 | 35/166 | 37/162
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP03-36 (0.15% Solution) (N=161) | MP03-33 (0.10% Solution) (N=166) | Placebo (N=162)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8) | 5 (5)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
dysgeusia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 1 (1)
uri (Infections and infestations) | 4 (4) | 4 (4) | 3 (3)
sneezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
pyrexia (General disorders) | 2 (2) | 2 (2) | 3 (3)
abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
nasopharynigitis (Infections and infestations) | 1 (1) | 5 (5) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 3 (3) | 4 (4)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5)
otitis media (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
pharyngitis streptoccal (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No